CLINICAL TRIAL: NCT07191054
Title: Prospective Trial Of Patient Outcomes and PALS Sepsis Guideline Adherence In Patients Fluid Resuscitated With The LifeFlow® Rapid Infuser Compared To Traditional Methods
Brief Title: LifeFlow Sepsis Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started, no enrollments.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-070
Record Dates: First submitted 2019-04-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Life Flow (Experimental): Patients concerning for severe sepsis will receive fluid resuscitation using the LifeFlow rapid infuser
  Interventions: Device: LifeFlow Rapid infuser
- Push-Pull (Active Comparator): Patients concerning for severe sepsis will receive fluid resuscitation using the standard push/pull technique
  Interventions: Device: Push Pull

INTERVENTIONS:
Device: LifeFlow Rapid infuser — Use of rapid infuser to fluid resuscitate
  Arms: Life Flow
Device: Push Pull — Use of Push Pull syringe technique to fluid resuscitate
  Arms: Push-Pull

SUMMARY:
This is a prospective, comparative, blinded, randomized study to prove the safety, efficacy and ease of use of the LifeFlow® device in pediatric patients presenting to an emergency department with concern for sepsis. This study will include 600 patients, 300 will receive the LifeFlow® device to deliver intravenous fluids while another 300 patients will receive the conventional push/pull method.

ELIGIBILITY:
Inclusion Criteria:

* Less than 19 years old
* Trigger the Best Practice Alert in triage
* Treating physician elects to do the full sepsis bundle.

Exclusion Criteria:

* Less than 20kg in weight
* Patients on diuretics for cardiac or renal conditions
* Patients who cannot communicate in either English or Spanish

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Time To first bolus completion | 20 Minutes
Time to third bolus completion | 60 Minutes
Time to hospital admission | 24 hours
  Time from presentation to the ER until admission to the hospital
Nursing satisfaction | 1 day
  Likert scale of satisfaction with style of fluid administration used. From not satisfied to extremely satisfied.

SECONDARY OUTCOMES:
Hospital Length of Stay | Days
ICU days | Days
Vasoactive medication use | 1 day
  Will measure whether vasoactive medications are used or not used
Morbidity and Mortality | 1 day
  rate of morbidity and mortality per 100 subjects in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No